CLINICAL TRIAL: NCT06739070
Title: Comparison Between Calisthenics and Plyometrics on Reducing Risk of Musculoskeletal Injuries Among School Going Children
Brief Title: Comparison Between Calisthenics and Plyometrics on School Going Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Riphah/RCRAHS-01924
Record Dates: First submitted 2024-10-23; First posted 2024-12-18 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Risk of MSK Injuries.; calisthenics; Plyometrics; school going children; functional movement screening; Deep Squat; Rotary stability; Shoulder Mobility; Trunk Pushups; Incline Lunges
MeSH Terms: interventions — Plyometric Exercise; Gymnastics; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calisthenics (Experimental): Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes. Session would be of 8 minutes in which 1 minutes exercise and 1 minute rest is there. Exercise include bunny jumps, bear crawls , crab walk and mad cat and 9 minutes cool down period. This protocol would be follow up to 8 weeks.
  Interventions: Other: Calisthenics
- Plyometric (Experimental): Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Interventions: Other: Plyometric
- Control (Other): compare with other groups
  Interventions: Other: Control group (no intervention)

INTERVENTIONS:
Other: Plyometric — Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Other Names: Group B
  Arms: Plyometric
Other: Calisthenics — Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Other Names: Group A
  Arms: Calisthenics
Other: Control group (no intervention) — In control group no intervention would be given. Initial test would be performed at 4th and 8th week and then results would be compared with experimental group.
  Other Names: Group C
  Arms: Control

SUMMARY:
Based on the provided document, here is a brief summary

The goal of this clinical trial is to compare the effects of calisthenics and plyometric exercises on reducing risk of MSK injuries among school-going children. The main questions it aims to answer are:

* Will calisthenics exercises have a better effect on reducing risk of MSK injuries compared to plyometric exercises in school-going children?
* How do these exercise interventions impact functional movements, and musculoskeletal pain improvements in children?

Researchers will compare a calisthenics exercise group, a plyometric exercise group, and a control group (no intervention) to see if there are differences in reducing risk of MSK injuries outcomes.

Participants will:

* Be male school-going children aged 8-12 years.
* Be randomly assigned to one of three groups: calisthenics, plyometric, or control.
* Complete baseline assessments of MSK (Functional Movement Screening and pain).
* Participate in their assigned exercise program 3 times per week for 8 weeks (exercise groups only).
* Complete follow-up assessments of MSK (Functional Movement Screening and pain) at 4 weeks and 8 weeks.
* Perform tests for functional movement screening and MSK assessment.

DETAILED DESCRIPTION:
Title: Comparison of Calisthenics and Plyometric Exercises on reducing risk of MSK Injuries Among School-Going Children.

This research study, conducted by Raees Fatima at Riphah International University in Islamabad, aims to investigate how different types of exercise affect cognitive abilities in children. Specifically, it compares the effects of calisthenics (bodyweight exercises) and plyometrics (jump training) on reducing risk of MSK Injuries in school-going children.

Key Details:

* Participants: Male school-going children aged 8-12 years
* Duration: 8 weeks
* Location: Public and private schools in Islamabad, Pakistan

The study will involve three groups:

1. Calisthenics group: Performing bodyweight exercises
2. Plyometric group: Engaging in jumping and explosive movement exercises
3. Control group: No specific exercise intervention

Both exercise groups will participate in supervised sessions three times per week. The exercises are designed to be age-appropriate and safe for children.

Measurements:

Researchers will assess various aspects of executive function using standardized tests:

- TNMQ'S FMS These assessments will be conducted at the beginning of the study, at 4 weeks, and at 8 weeks to track changes over time.

Significance:

This study is important because it could provide valuable insights into how different types of exercise reduces risk of MSK Injuries. The results could inform physical education programs in schools and help parents and educators make informed decisions about children's physical activities.

Ethical Considerations:

The study has been approved by the university's ethics review board. Participation is voluntary, and parents must provide informed consent. All data will be kept confidential and coded to protect participants' identities.

Expected Outcomes:

The researchers hypothesize that calisthenics exercises may have a more significant positive effect on reducing risk of MSK Injuries compared to plyometric exercises. However, both exercise types are expected to show improvements compared to the control group.

This research contributes to the growing field of exercise neuroscience and could have practical implications for child development, education, and public health policies related to physical activity in schools.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Male School Going Children (8-12 Years Of Age)
* Normal BMI of School Going Children
* No Recent Musculoskeletal Injury from last month.
* Not Actively Engaged In Other Sports

Exclusion Criteria

* Children with any mental or physical disability.
* Children with acute illness or fracture
* Active Inflammation or infections
* Any physical deformity

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — male participants
Enrollment: 99 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Deep Squat (FMS) | 8 weeks
  The mechanics of a deep squat include:
  Starting position Stand with feet shoulder-width apart and toes turned out slightly. knees should be straight.
  Lowering Bend hips and knees simultaneously, keeping back straight and chest up. knees should travel forward over toes, and hips should travel backward.
  Lowest position Hips should be as low as can go, ideally below knees. Pelvis should be in a neutral position, aligned with shins.
  Rising Push through heels and drive hips upward. Engage core and glutes to return to the starting position.
  Joint mobility Deep squats require a lot of mobility in your hips, knees, ankles, and lumbar spine.
  Trunk position Maintaining a neutral spine position allows for better control of compressive loads and shear forces.
Hurdle Step (FMS) | 8 weeks
  The mechanics of a hurdle step include:
  Takeoff The takeoff foot loses contact with the ground, and the hip flexes and abducts. The heel of the trail leg folds near the buttocks, and angular momentum transfers to the lower leg.
  Trail leg The knee of the trail leg should remain higher than the ankle. The foot should be everted to allow clearance.
  Upper body The lead arm sweeps wider to counter the trail leg's wider path. Landing The trail leg moves downward to resume sprinting. The lower leg should remain aligned as the hip drives it toward the ground.
  Displacement The body should move significantly beyond the takeoff foot before flight. Displacement should start in the core of the body, not the limbs.
  Body lean A forward lean may be needed to aid clearance, but it shouldn't disturb postural alignment.
  Lead leg hip The lead leg hip should flex and extend rapidly to avoid hitting the hurdle with the lead foot.
Incline Lunge (FMS) | 8 weeks
  Here are some mechanics for performing incline lunges:
  Form: Start with a box or incline that's 4-8 inches high. Step forward with front leg until knee is about 90 degrees.
  Glutes: Incline lunges target glutes more than a regular walking lunge. Hips: Push hips back when bend, and then push them forward when stand. Shoulders and chest: Keep shoulders back and chest lifted. Balance: If using a dumbbell, hold it in opposite hand to help with balance. Feet: Make sure feet are far enough apart so that your front knee stays over your ankle.
  Back knee: Drop back knee down. Motion: Do an up-and-down motion, don't lean forward. Legs: Incline lunges work on quads, glutes, and hamstrings.
Shoulder Mobility (FMS) | 8 weeks
  To do this test, stand up straight and make a fist with each hand. Place one fist on opposite shoulder and the other behind back on the same side. Try to bring elbows as close as possible without moving your torso.
Impingement Clearing Test (FMS) | 8 weeks
  The shoulder clearing test is a pain-free procedure that checks for shoulder impingement:
  Reach one hand across body and place it against opposite shoulder. Apply inward pressure while slowly raising elbow. Repeat on the other side.
Active Straight Leg Raise (FMS) | 8 weeks
  The subject is instructed to raise one leg, then the other, without bending the knee, until the heel is 20 cm above the table.
  The subject is asked to hold the leg elevated for about 10 seconds. The subject is asked to rate the difficulty of the test on a scale of 0 to 5. The subject is asked if one leg feels heavier than the other or if there is any pain.
Trunk Stability Pushup (FMS) | 8 weeks
  Lie on stomach with hands shoulder-width apart Position thumbs in line with forehead if male, or chin if female Tighten core and raise body off the ground in one line Try to arch back as little as possible Push body up into a push-up position as one unit Ensure there's no lag in spine.
Press up Clearing Test | 8 weeks
  The press-up clearing test is a part of the Functional Movement Screen (FMS) that assesses pain response and is used to identify individuals at risk of injury:
  Position The participant lies on stomach with hands placed shoulder-width apart and palms down.
  Instructions The participant should raise toes toward shins and place them on the ground, extend their knees, and maintain a rigid torso.
  Execution The participant should press their chest off the floor by extending their elbows, arching their back as much as possible, and keeping their hips in contact with the floor.
  Scoring If the participant experiences pain at any point during the test, they receive a score of zero and the test is terminated. The painful area should be noted.
Rotary Stability (FMS) | 8 Weeks
  The procedure involves the following steps:
  Get on all fours with your hands and knees on a board, with arms and thighs vertical and toes resting on the floor.
  Simultaneously reach right arm forward and extend your right leg backward. Retract elbow and right knee until they touch directly over the board. Repeat the movement at least twice without touching the floor with arm or leg. Repeat the test on the other side. If can't complete the movement within three attempts, can try a modified diagonal flexion and extension lift.
  The test administrator will assess performance based on whether hand and leg clear the floor by about 6 inches (15 cm) and whether make contact with the floor while performing the repetitions.
Posterior Rocking Clearing Test (FMS) | 8 weeks
  Posterior rocking clearing test is performed:
  Assume a quadruped position Rock back and touch the buttocks to the heels and the chest to the thighs Keep the hands in front of the body and reach out as far as possible
  The FMS is a series of seven tests that evaluate fundamental movement patterns. The tests are designed to identify movements that increase the risk of injury and insufficient movement that reduces performance. The FMS uses a four-point scale to score each test:
  3: The movement task was performed perfectly without compensations 2: The task was completed with compensatory movements
  1: The participant was unable to perform the movement as required 0: The participant felt pain during the movement task

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, Phd, Principal Investigator — Riphah International University
Locations (1):
- Different Schools, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No